CLINICAL TRIAL: NCT01626027
Title: Depression Care for Hospitalized Coronary Heart Disease Patients: Bridging the Gap Between Guidelines and Reality
Brief Title: Depression Care for Hospitalized Coronary Heart Disease Patients: Prospective Cohort Study
Acronym: CDCare
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Jacqueline Müller-Nordhorn, Professor, Charite University, Berlin, Germany
Other Study IDs: 01GY1154
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Heart Disease; Depression
Keywords: Coronary Heart Disease; Depression; Health Care Services
MeSH Terms: conditions — Coronary Disease; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this prospective, observational study are to assess the current use of depression care in Coronary Heart Disease (CHD) patients, and to provide estimates for the resources needed to implement guideline-oriented depression health care acceptable to CHD patients with comorbid depression.

DETAILED DESCRIPTION:
In patients with established CHD, unipolar depression is up to three times more prevalent than in the general population and increases the risk for coronary events and mortality, higher health care consumption and decreased quality of life. Most hospitals in Germany have a unique infrastructure of psychiatric, psychosomatic and psychosocial services for CHD patients (psychiatric/psychosomatic consultation liaison services and a wide network of inpatient or outpatient cardiac rehabilitation centers). However, as of today, little is known about the current use and acceptability of depression health care from the perspective of CHD patients.

This project has two main aims:

1. to assess the current use of depression care in CHD patients who are hospitalized or receive ambulatory care at a cardiology clinic
2. to provide estimates for the resources needed to implement guideline-oriented depression health care acceptable to CHD patients with comorbid depression.

Specifically, the investigators will assess

* rates of and satisfaction with depression health care use in hospitalized CHD patients within one year after hospitalization
* perceived need for depression care and patient preferences for different types, settings and providers of these services
* correlates of depression health care use and patient preferences
* the amount of patients in need for depression health care according to existing recommendations

The secondary objective is to assess direct and indirect costs associated with depressive symptoms and depression care use across 1 year (as indicated by quality of life, event-free survival, productivity, and health care costs).

ELIGIBILITY:
Inclusion Criteria:

* chronic CHD (confirmed by a clinician)

Exclusion Criteria:

* chart-documented dementia disorder
* cognitive impairment
* life expectancy < 1 year
* unavailability for follow-up
* insufficient proficiency in German or Turkish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed Coronary Heart Disease (CHD) hospitalized in the coronary care units of 2 University hospitals in Germany. Additionally, starting August 2012, patients with confirmed CHD who receive ambulatory care at one of the cardiology clinics will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1265 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in depression care during the 12 months after hospitalization | Baseline and within one year after hospitalization
  Assessed via questionnaire (self-reported psychotherapy for depression and / or antidepressant medication and / or other treatment) at baseline, 1month, 6 month and 12 months Additionally, antidepressant medication prescription will be assessed at baseline via chart review (antidepressant medication at admission and discharge)

SECONDARY OUTCOMES:
Percentage of participants reporting current utilization of mental health care and satisfaction with mental health care | Baseline and within one year after hospitalization
  Current mental health care utilization is assessed via questionnaire with a single item ("yes or no").
  Satisfaction with current mental health care is assessed via questionnaire with a single continuous rating item (ranging from "very satisfied to not at all satisfied") at baseline and all follow-up assessments (1mo, 6mo and 12months)
Patient preferences for different providers and settings of mental health care services, as indicated by the percentage of patients who indicate actual receipt of or potential willingness to receive mental health care by specific providers and settings | Baseline and within one year after hospitalization
  Assessed via questionnaire with at baseline and all follow-up assessments (1mo, 6mo and 12months). A list of mental health care providers (e.g., general practitioner, psychotherapist, psychiatrist, ...) is provided and for each, patients are asked to indicated whether they currently receive mental health care from any provider and if not, if they would be willing to reciev mentral health care by that provider, should they ever be in need (answer options "yes, maybe, no").
Percentage of patients in need for depression health care according to existing recommendations | Baseline and within one year after hospitalization
  Baseline: Percentage of patients with a current Major Depressive Episode as assessed via the Composite International Diagnostic Interview (CIDI).
  6 months assessment: percentage of patients with a current Major Depressive Episode as assessed via the Composite International Diagnostic Interview (CIDI) - this will only be conducted in a subsample of 300 consecutive participants.
  Follow-up assessments: percentage of patients with persistently elevated depressive symptoms as indicated by a score of >=10 on the Patient Health Questionnaire (PHQ-9) at baseline and the follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Müller-Nordhorn, MD, DPH, Principal Investigator — Charité Universitätsmedizin
Locations (1):
- Medizinische Klinik m. Schwerpunkt Kardiologie, Charité Universitätsmedizin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided